CLINICAL TRIAL: NCT07270250
Title: Impact of Dry vs Humidified Culture Conditions on Blastocyst Development and Aneuploidy: A Time-lapse Sibling Oocyte Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, leroy vas, Embryologist, ART Fertility Clinics LLC
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2504-ABU-013-LV
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Incubator Stay; Total Blastulation; Blastocyst Quality; Biopsy Rate; Fertilization Rate; Ploidy Rate; ICSI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Chamber of Geri (Other)
  Interventions: Device: K- system incubator
- Humidified Chamber of Geri (Other)
  Interventions: Device: K- system incubator

INTERVENTIONS:
Device: K- system incubator — Following oocyte retrieval, collected oocytes will be incubated in Global Total for Fertilization within a K-Systems incubator until the time of denudation and intracytoplasmic sperm injection (ICSI). All mature (MII) oocytes will undergo ICSI at 39-41 hours post-trigger. After insemination, sibling oocytes will be divided as equally as possible and randomly allocated into two separate Geri incubator chambers: Group 1 will be cultured in the dry chamber, and Group 2 will be cultured in the humidified chamber. A predefined randomization list will determine allocation, including cases with an uneven number of oocytes, where the additional oocyte will be assigned according to the list. Both groups will use Global TotalR (GT, CooperSurgical) single-step medium. Embryo culture will be carried out in continuous culture conditions until the blastocyst stage, following the manufacturer's GT protocol, with no Day 3 media refreshment. To minimize procedural variability, one operator will ideally

SUMMARY:
IVF incubators are essential for maintaining the micro-environment required for embryo development. Incubator technology has progressed from early humidified box systems to benchtop and now time-lapse platforms, driving the development of dry incubator chambers. Both humidified and dry systems have specific pros and cons. Evidence to date suggests that humidified chambers may support better blastocyst development in certain "no-refresh" continuous culture conditions, but current data are limited and study designs remain weak. This study aims to compare sibling oocytes cultured in dry versus humidified chambers within a GERI time-lapse incubator under continuous culture conditions, assessing effects on viability and developmental outcomes. Findings may inform optimal incubation strategies to improve IVF success rates while supporting uninterrupted workflows and potentially improving cost-benefit efficiency in the IVF laboratory.

ELIGIBILITY:
Inclusion Criteria:

* PGT-A cycles with more than at least 4 mature oocytes
* ICSI
* maternal age 18- 43 years old
* PGT-A intended cycles with trophectoderm biopsies on day 5 /6/7
* patients with more than 8 oocytes expected for ICSI
* BMI <35
* fresh and frozen ejaculated sperm

Exclusion Criteria:

* PGT-M /PGT-SR cycles
* fresh and frozen testicular sperm
* IVF insemination
* previous history of fertilization failure

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Day 5 blastulation versus total blastulation | Day 5 post-insemination
  Day 5 blastulation versus total blastulation refers to comparing the proportion of embryos that reach the blastocyst stage specifically by Day 5 against the overall number of embryos that eventually form blastocysts
Blastocyst quality at time of biopsy based on modified Gardner's criteria. | Day 5 post-insemination
  Blastocyst quality at the time of biopsy will be assessed using the modified Gardner's grading system, which evaluates three key components of the blastocyst: the degree of expansion, the quality of the inner cell mass (ICM), and the quality of the trophectoderm (TE). This standardized scoring allows objective comparison of embryo morphology and developmental competence at the moment of trophectoderm biopsy.

SECONDARY OUTCOMES:
Total blastulation rates per MII and 2PN. | Day 5 post-insemination
  Total blastulation rates per MII and per 2PN refer to the proportion of inseminated mature oocytes (MII) and normally fertilized zygotes (2PN) that successfully develop into blastocysts, regardless of whether they reach this stage on Day 5 or Day 6. This measurement reflects the overall efficiency of embryo development from both the point of maturation and normal fertilization.
Ploidy rate/biopsy and types of aneuploidies (segmental and mosaic) | Day 5 post-insemination
  Ploidy rate per biopsy refers to the proportion of biopsied blastocysts that return a euploid, aneuploid, mosaic or segmental result after PGT-A testing. This includes reporting the distribution of chromosomal abnormalities identified, distinguishing between full aneuploidies (whole chromosome gain or loss), segmental aneuploidies (partial chromosome changes) and mosaic patterns (mixed normal and abnormal cell lines). This outcome reflects the chromosomal competence of embryos generated under each culture condition.
Blastocyst utilization rate | 30 days
  Blastocyst utilization rate refers to the proportion of blastocysts that are suitable for clinical use-meaning those that are either transferred, frozen for future use, or biopsied for PGT-A.
Rate of day 5 biopsy | Day 5 post-insemination
  Rate of Day 5 biopsy refers to the proportion of blastocysts that reach the biopsy stage specifically on Day 5, relative to the total number of blastocysts biopsied.

CONTACTS AND LOCATIONS:
Overall Officials: BARBARA LAWRENZ, PhD, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
upon request

REFERENCES:
- [Result] Bartolacci A, Borini A, Cimadomo D, Fabozzi G, Maggiulli R, Lagalla C, Pignataro D, dell'Aquila M, Parodi F, Patria G, Zaca C, Ubaldi FM, Rienzi L, Coticchio G. Humidified atmosphere in a time-lapse embryo culture system does not improve ongoing pregnancy rate: a retrospective propensity score model study derived from 496 first ICSI cycles. J Assist Reprod Genet. 2023 Jun;40(6):1429-1435. doi: 10.1007/s10815-023-02818-8. Epub 2023 May 3. PMID 37133689
- [Result] Ueno S, Ito M, Shimazaki K, Okimura T, Uchiyama K, Yabuuchi A, Kato K. Comparison of Embryo and Clinical Outcomes in Different Types of Incubator Between Two Different Embryo Culture Systems. Reprod Sci. 2021 Aug;28(8):2301-2309. doi: 10.1007/s43032-021-00504-7. Epub 2021 Mar 9. PMID 33751461
- [Result] Fawzy M, AbdelRahman MY, Zidan MH, Abdel Hafez FF, Abdelghafar H, Al-Inany H, Bedaiwy MA. Humid versus dry incubator: a prospective, randomized, controlled trial. Fertil Steril. 2017 Aug;108(2):277-283. doi: 10.1016/j.fertnstert.2017.05.036. Epub 2017 Jun 23. PMID 28651960
- [Result] Chi HJ, Park JS, Yoo CS, Kwak SJ, Son HJ, Kim SG, Sim CH, Lee KH, Koo DB. Effect of evaporation-induced osmotic changes in culture media in a dry-type incubator on clinical outcomes in in vitro fertilization-embryo transfer cycles. Clin Exp Reprod Med. 2020 Dec;47(4):284-292. doi: 10.5653/cerm.2020.03552. Epub 2020 Nov 23. PMID 33227188
- [Result] Cheredath A, Uppangala S, Asampille G, Lakshmi R V, Joseph D, Raval K, Gowda G A N, Kalthur G, Adiga SK. Duration of dry and humidified incubation of single-step embryo culture medium and oxygen tension during sham culture do not alter medium composition. F1000Res. 2022 Feb 28;11:242. doi: 10.12688/f1000research.109895.4. eCollection 2022. PMID 35811802
- [Result] Castillo CM, Harper J, Roberts SA, O'Neill HC, Johnstone ED, Brison DR. The impact of selected embryo culture conditions on ART treatment cycle outcomes: a UK national study. Hum Reprod Open. 2020 Feb 10;2020(1):hoz031. doi: 10.1093/hropen/hoz031. eCollection 2020. PMID 32083189